CLINICAL TRIAL: NCT00741871
Title: A Phase 1 Study of SB1518 for the Treatment of Advanced Lymphoid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SB1518-2007-002
Record Dates: First submitted 2008-08-22; First posted 2008-08-26 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Lymphoma, Malignant; Hodgkin's Lymphoma; B Cell Lymphoma
Keywords: Lymphoid malignancies; Hodgkin's Lymphoma; Diffuse large B cell lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB1518 — SB1518 taken orally daily for 28 consecutive days in a 28 day cycle

SUMMARY:
This is a Phase 1 dose escalation study to determine the maximum tolerated dose and the dose limiting toxicities of SB1518 when given alone once daily by mouth to subjects with advanced lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically documented diagnosis of a lymphoid malignancy as defined in the World Health Organization (WHO) classification scheme except for those listed in Exclusion Criteria
* Subject must have received at least 2 prior regimens for their lymphoid malignancy, one of which was an anthracycline-containing combination regimen and have shown disease relapse or did not respond to the prior regimen
* Subjects with classic HL or diffuse large B cell lymphoma must have failed, refused or are ineligible to receive stem cell transplant
* Subjects must have measurable lesions (at least one target lesion measuring 2cm in diameter) by computerized tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* All men of reproductive potential and women of child-bearing potential must agree to practice effective contraception during the entire study period and for one month after the last study treatment unless documentation of infertility exists. Additionally, women of child-bearing potential must have a negative pregnancy test within 14 days prior to the first dose of study drug
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

* Post-Transplant Lymphoproliferative Disease (PTLD), Burkitt's lymphoma, Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, multiple myeloma, or HIV-associated lymphoma
* History of or active Central Nervous System (CNS) malignancy
* Have undergone allogeneic stem cell transplant and were treated with immunosuppressing agent within the past 6 months
* Active Graft-versus-host disease (GVHD)
* Uncontrolled inter-current illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as judged by treating physician. Subjects receiving antibiotics for infections that are under control may be included in the study
* Concurrent malignancy, except those subjects with early stage squamous cell carcinoma of the skin, basal cell carcinoma of the skin, or cervical intraepithelial neoplasia are eligible for the study
* Known HIV-positive (such subjects are at increased risk of lethal infections when treated with potentially marrow-suppressive therapy)
* Known active Hepatitis A, B or C
* Women who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To establish the maximum tolerated dose of SB1518 as a single agent when administered orally daily in subjects with advanced lymphoid malignancies. | Throughout the study

SECONDARY OUTCOMES:
To assess the safety and tolerability of SB1518, administered orally once daily in subjects with advanced lymphoid malignancies. | Throughout the study
To assess the pharmacokinetic and pharmacodynamic profile of SB1518. | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Anas Younes, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Younes A, Romaguera J, Fanale M, McLaughlin P, Hagemeister F, Copeland A, Neelapu S, Kwak L, Shah J, de Castro Faria S, Hart S, Wood J, Jayaraman R, Ethirajulu K, Zhu J. Phase I study of a novel oral Janus kinase 2 inhibitor, SB1518, in patients with relapsed lymphoma: evidence of clinical and biologic activity in multiple lymphoma subtypes. J Clin Oncol. 2012 Nov 20;30(33):4161-7. doi: 10.1200/JCO.2012.42.5223. Epub 2012 Sep 10. PMID 22965964